CLINICAL TRIAL: NCT04340375
Title: A Clinical Study to Evaluate the Anti-pollution Effects of AP Green Tea Extracts in Subjects With Discomforts Related to the Respiratory System by Prolonged Exposure to Particulate Matter in Air Pollution
Brief Title: Anti-pollution Effects of AP Green Tea Extracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AP-R-2018-01
Record Dates: First submitted 2020-03-31; First posted 2020-04-09 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Conditions Due to Unspecified External Agent
Keywords: Anti-pollution; green tea extracts

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AP green tea extracts (Experimental): 8 weeks
  Interventions: Dietary Supplement: AP green tea extracts

INTERVENTIONS:
Dietary Supplement: AP green tea extracts — AP green tea extracts

SUMMARY:
The objective of this clinical trial is to evaluate the anti-pollution effects of AP green tea extracts in subjects with discomforts related to the respiratory system by prolonged exposure to particulate matter in air pollution

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 19 years or over
* Subjects with discomforts related to the respiratory system by prolonged exposure to particulate matter in air pollution
* Subjects who voluntarily decide to participate in this clinical study and sign the informed consent form on their own or through their representatives

Exclusion Criteria:

* At the screening visit, subjects who were diagnosed with acute or chronic respiratory disease and undergoing medication.
* Subjects who were diagnosed with ventricular associated disease, unstable and uncontrolled chronic medical disease, or active malignant tumor and undergoing medication within 4 weeks prior to the first administration of the investigational product
* Subjects who show a level of ALT/AST of 2 times or more the upper limit of normal as a result of a screening test and have acute or chronic hepatitis or known liver cirrhosis
* In addition to the above, subjects who are determined to be ineligible to participate in the clinical study according to the investigator's medical opinion

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test | 4 weeks
  Improvement in pulmonary function test
Pulmonary function test | 8 weeks
  Improvement in pulmonary function test
Respiratory health survey | 4 weeks
  Patients' self evaluation of COPD Assessment Test
Respiratory health survey | 8 weeks
  Patients' self evaluation of COPD Assessment Test
Biomarkers | 4 weeks
  Blood concentration of biomarkers (Inflammatory cytokines)
Biomarkers | 8 weeks
  Blood concentration of biomarkers (Inflammatory cytokines)
Heavy metals | 4 weeks
  Blood concentration of heavy metals
Heavy metals | 8 weeks
  Blood concentration of heavy metals

SECONDARY OUTCOMES:
Bronchial assessment | 4 weeks
  Patients' self evaluation of Bronchiectasis Health Questionnaire
Bronchial assessment | 8 weeks
  Patients' self evaluation of Bronchiectasis Health Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No